CLINICAL TRIAL: NCT03171259
Title: SCOPE CLI (Shifting Care and Outcomes for Patients With Endangered Limbs- Critical Limb Ischemia)
Brief Title: SCOPE CLI (Shifting Care and Outcomes for Patients With Endangered Limbs - Critical Limb Ischemia)
Acronym: SCOPE CLI
Status: Completed | Type: Observational
Sponsor: Saint Luke's Health System (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-054
Record Dates: First submitted 2017-05-23; First posted 2017-05-31 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: care as usual — The investigators will be following patients with critical limb ischemia and documenting the usual care that the participants receive.

SUMMARY:
Given the importance of understanding CLI patients' outcomes and existing gaps in knowledge, there is a pressing need to collect observational data on treatment patterns, adherence to performance measures, and outcomes that are relevant to patients and clinicians. To address this need, the current study will pilot test the research infrastructure and data elements needed to build a larger, national study collecting of the CLI population. It will also provide much-needed preliminary information to identify areas of action that can be targeted in quality improvement programs for this population. Most importantly, it will provide data on health status outcomes in patients with CLI, as a function of individual patient characteristics (demographics, socio-economic and clinical background) and the treatments that patients have undergone. The PORTRAIT-CLI study will also be well equipped to identify potential disparities in the provision of care and patients' outcomes as a function of patient's characteristics.

ELIGIBILITY:
Inclusion Criteria:

All race/ethnicity categories, English or Spanish speaking, men and women

* Age ≥18 years
* Patients presenting with Rutherford Classification 4 (ischemic rest pain), or Rutherford Classification 5 (minor tissue loss: non-healing ulcer, focal gangrene with diffuse pedal ischemia), or Rutherford Classification 6 (major tissue loss: extending above transmetatarsal level, functional foot no longer salvageable) at specialty clinics will prospectively be screened, regardless of whether the patient undergoes endovascular, bypass, amputation, and/or medical therapy.
* Diagnosis is supported by any of the following hemodynamic parameters (assessed pre- procedurally): Ankle pressure lower than 70 mmHg; Toe pressure lower than 50 mmHg or evidence of ischemia by transcutaneous oxygen measurement (tcpO2) <40 or a skin perfusion pressure (SPP) <40 or angiographic evidence of significant vascular disease

Exclusion Criteria:

* No other prior surgical or vascular interventions within 2 weeks before and/or planned 30 days after the enrollment
* Acute limb ischemia
* Unable to provide written informed consent
* Currently a prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Project coordinators at each recruitment site will have direct access to the PAD clinic schedules and will be prospectively screening from that list. A screening form with limited demographic information will be completed for all patients with a diagnosis of CLI supported by any of the following hemodynamic parameters (assessed pre-procedurally): Ankle pressure lower than 70 mmHg; Toe pressure lower than 50 mmHg or evidence of ischemia by transcutaneous oxygen measurement (tcpO2) <40 or a skin perfusion pressure (SPP) <40 or angiographic evidence of significant vascular disease.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
CLI-specific health status | 12 months
  Peripheral Artery Questionnaire-CLI version

SECONDARY OUTCOMES:
Freedom from major amputation or major reintervention | 12 months
  Freedom from major amputation or major peripheral vascular reintervention (surgical or angioplasty)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Smolderen, PhD, Principal Investigator — University of Missouri Kansas City; Saint Luke's Hospital
Locations (2):
- United States (2):
  - Yale New Haven Hospital, New Haven, Connecticut
  - University Hospitals Cleveland, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bradbury AW, Adam DJ, Bell J, Forbes JF, Fowkes FG, Gillespie I, Ruckley CV, Raab GM; BASIL trial Participants. Bypass versus Angioplasty in Severe Ischaemia of the Leg (BASIL) trial: Analysis of amputation free and overall survival by treatment received. J Vasc Surg. 2010 May;51(5 Suppl):18S-31S. doi: 10.1016/j.jvs.2010.01.074. PMID 20435259
- [Background] Spertus J, Jones P, Poler S, Rocha-Singh K. The peripheral artery questionnaire: a new disease-specific health status measure for patients with peripheral arterial disease. Am Heart J. 2004 Feb;147(2):301-8. doi: 10.1016/j.ahj.2003.08.001. PMID 14760329
- [Result] Adam DJ, Beard JD, Cleveland T, Bell J, Bradbury AW, Forbes JF, Fowkes FG, Gillepsie I, Ruckley CV, Raab G, Storkey H; BASIL trial participants. Bypass versus angioplasty in severe ischaemia of the leg (BASIL): multicentre, randomised controlled trial. Lancet. 2005 Dec 3;366(9501):1925-34. doi: 10.1016/S0140-6736(05)67704-5. PMID 16325694